CLINICAL TRIAL: NCT02005770
Title: Does Anesthesia Technique Affect the Presence of Circulating Tumor Cells in Primary Breast Carcinoma? A Randomised Controlled Trial.
Brief Title: Anesthesia and Circulating Tumor Cells in Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-0408
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Female Breast Carcinoma
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Experimental): General anesthesia using Sevoflurane
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): General anesthesia using propofol TCI
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Sevoflurane
Drug: Propofol
  Arms: Propofol

SUMMARY:
Serious concern about the role of anesthesia in tumor recurrence has considerably risen over years, but the lack of surrogate markers for tumor spreading made trials addressing this issue difficult to realize. In breast cancer patients CTC positivity has been recently recognized as an independent prognostic factor. In this respect, we postulated that in a first step changes in the number of CTC after general anesthesia would help to determine the effect of anesthesia on this tumor marker.

DETAILED DESCRIPTION:
Patients with primary breast cancer will be randomized to either propofol or sevoflurane anesthesia for curative surgery. CTC will be determined in the pre- as well as postoperative phase and the kinetic of CTC in the two groups will be compared.

ELIGIBILITY:
Inclusion criteria: > Female

* Age 18 to 85
* ASA I-III
* Primary breast cancer (TNM stage = T1-3, N0-2, M0)
* Primary surgery
* Written informed consent

Exclusion criteria:

* Metastatic breast cancer
* Other than primary surgery (recurrence, reconstruction)
* Pre-operative chemotherapy or radiotherapy
* Auto-immune disease, HIV, other active cancer, age>85, ASA IV or V
* Concomitant regional anesthesia
* Chronic opioids medication
* Any systemic immunosuppressive therapy
* Known hypersensitivity or suspected allergy to propofol, soya or egg proteins
* Known hypersensitivity to volatile anesthetics (malignant hyperthermia)
* Pregnancy
* Breast feeding
* Non German-speaking patients
* Enrollment in any other clinical trial during the course of this trial, 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number of CTC before and after administration of anesthetics | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof MD, Principal Investigator — University Hospital Zurich, Institute of Anesthesiology
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Institute of Anesthesiology, Zurich, Canton of Zurich
  - Institute of Physicians for Anesthesia and Intensive Care Klinik Hirslanden, Zurich

REFERENCES:
- [Derived] Hovaguimian F, Braun J, Z'graggen BR, Schlapfer M, Dumrese C, Ewald C, Dedes KJ, Fink D, Rolli U, Seeberger M, Tausch C, Papassotiropoulos B, Puhan MA, Beck-Schimmer B. Anesthesia and Circulating Tumor Cells in Primary Breast Cancer Patients: A Randomized Controlled Trial. Anesthesiology. 2020 Sep;133(3):548-558. doi: 10.1097/ALN.0000000000003409. PMID 32568845

DOCUMENTS (1):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02005770/Prot_000.pdf